CLINICAL TRIAL: NCT05110183
Title: Opto-Electrical Cochlear Implants
Acronym: oCI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Central DuPage Hospital (Other); University of Miami (Other); University of Missouri-Columbia (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU00209027; R01DC018666 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss
Keywords: deaf; neural stimulation with light; cochlear implant
MeSH Terms: conditions — Hearing Loss | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- electrical and optical hybrid stimulation stimulation (Experimental): Patients with large tumors of the skull base, requiring a translabyrinthine craniotomy with sacrifice of their cochlea and vestibular system during the tumor resection may participate. A recording electrode will be placed on the round window, a cochleostomy will be created, and different Light delivery systems (LDSs) will be inserted into the cochlea. LDSs include angle polished optical fibers to determine the accuracy of the orientation of the radiation beam, and hybrid arrays of small optical sources and electrical contacts to evaluate electric-alone stimulation as a reference, and compare it to optic-alone and combined electrical and optical stimulation. Compound action potentials (CAPs) of the auditory nerve will be recorded.
  Interventions: Device: electrical stimulation; Other: optical stimulation; Other: combined optical and electrical stimulation

INTERVENTIONS:
Device: electrical stimulation — A cochlear implant electrode will be inserted through a cochleostomy into scala tympani of the cochlear basal turn. Custom software on a laptop computer will be used to control the delivery of a sequence of charge balanced current pules.
Other: optical stimulation — Optical fibers will be inserted through a cochleostomy into scala tympani of the cochlear basal turn. Custom software will be used to control the delivery of a sequence of charge balanced current pules.
Other: combined optical and electrical stimulation — A short hybrid array consisting of optical sources and electrical contacts will be inserted through a cochleostomy into scala tympani of the cochlear basal turn. Biphasic electrical current pulse and optical pulse delivery will be controlled in amplitude and timing by a computer.

SUMMARY:
Neural stimulation with photons has been proposed for a next generation of cochlear implants (CIs). The potential benefit of photonic over electrical stimulation is its spatially selective activation of small populations of spiral ganglion neurons (SGNs). Stimulating smaller neuron populations along the cochlea provides a larger number of independent channels to encode acoustic information. Hearing could therefore be restored at a higher fidelity and performance in noisy listening environments as well as music appreciation are likely to improve .

While it has been demonstrated that optical radiation evokes auditory responses in animal models, it is not clear whether the radiant exposures used in the animal experiments are sufficient to stimulate the auditory system of humans. The proposed tests are:

1. to demonstrate that light delivery systems (LDSs) can be inserted and oriented optimally in the human cochlea.
2. to show that the LDSs are able to deliver sufficient amount of energy to evoke a compound action potential of the auditory nerve.
3. to validate that the fluence rate (energy / target area) required for stimulation is below the maximal fluence rate, which damaged the cochlea in animal experiments.
4. to show that combined optical and electrical stimulation is able to significantly lower the threshold required for optical stimulation in humans.

The endpoints for the study are either the completion of the experiments proposed or the demonstration that not sufficient energy can be delivered safely in the human cochlea to develop an action potential.

DETAILED DESCRIPTION:
The patient is admitted to one of the participating clinical centers because of a brain tumor, which requires surgery to be removed. As discussed in detail with the treating surgeon, the tumor is large, and an approach will be used that accesses the tumor from the side through the temporal bone. This approach passes by the balance and hearing organ, and the partial or complete removal of the organ responsible for balance and hearing on this side is necessary. Participation in the study will extend the time of surgery by 30 minutes. There is no special preparation and no follow-up required for the study.

In this study, a cochlear implant system that uses light to stimulate the cochlea will be tested. It is a small light delivery system consisting of optical fibers and light sources the size of a human hair. This light delivery system will be inserted into the hearing organ, the cochlea before it is damaged or removed during the tumor surgery. After insertion into the cochlea, pulses of infrared light will be delivered to the cochlea, and auditory responses will be measured with a small electrode placed at the cochlea.

If possible, after completion of the measurements and during the continuation of the tumor surgery, the tissue of the hearing organ, which is typically destroyed through the drilling, will be harvested for histological evaluation.

ELIGIBILITY:
Inclusion Criteria:

Criterion for inclusion of a patient is the requirement of the translabyrinthine approach for tumor removal. The surgical approach is determined by the tumor size, the tumor location and the remaining hearing of the patient. Criteria for a translabyrinthine approach are:

1. the tumor grows in the pontine angle and the facial nerve is at risk for damage during the surgery because the tumor is already large and in close proximity of the facial nerve AND
2. the tumor is larger than 2.5 cm AND
3. Pure tone hearing thresholds are elevated by at least 50 dB AND
4. Speech discrimination scores are 50% or less

Exclusion Criteria:

* adults unable to consent.
* individuals who are not yet adults (infants, children, teenagers).
* pregnant women.
* prisoners.
* vulnerable populations

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Compound Action Potential (CAP) | 30 minutes
  Compound action potentials (CAPs) of the auditory nerve in response to electrical stimulation, optical stimulation, and combined optical and electrical stimulation will be recorded. Electrical stimulation alone is used to determine baseline cochlear function. Optical stimulation alone will then be used to determine a similar baseline for optical stimulation and test parameters such as optical pulse rate, pulse duration and radiant exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Claus-Peter Richter, MD, PhD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - University of Miami, Coral Gables, Florida
  - Central DuPage Hospital Association, Winfield, Illinois
  - University of Missouri, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At publication of the results.
Access Criteria: With the publication the study, de-identified data will be uploaded to a data repository and are accessible through figshare.com.
URL: http://figshare.com